CLINICAL TRIAL: NCT07171073
Title: Changes in Biosocial and Cognitive Functions and Quality of Life When Applying Different Smart Technologies in Stroke Patients During Early Rehabilitation
Brief Title: Smart Technologies in Early Post-Stroke Rehabilitation
Acronym: SMART-Stroke
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Erika Endzelyte (Other)
Collaborators: The Hospital of Lithuanian University of Health Sciences Kaunas Clinics (Unknown); Kulautuva Hospital of Rehabilitation (Unknown)
Responsible Party: Sponsor-Investigator, Erika Endzelyte, Researcher, Lithuanian University of Health Sciences
Organization: Lithuanian University of Health Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LSMU-2025-StrokeRehab
Record Dates: First submitted 2025-08-28; First posted 2025-09-12 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Stroke
Keywords: Stroke rehabilitation; Cognitive function; Quality of life; Smart technologies; Virtual reality; Brain-computer interface (BCI); Robot-assisted rehabilitation; Occupational therapy
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Outcome assessors will be blinded to group assignment; participants and care providers will be aware of the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- RecoveriX Group (Experimental): Stroke patients receiving interactive rehabilitation with the RecoveriX brain-computer interface (BCI) system.
  Duration: 6-7 weeks, in addition to conventional rehabilitation.
  Interventions: Device: RecoveriX
- Gloreha Aria Group (Experimental): Stroke patients receiving robotic-assisted therapy with the Gloreha Aria system.
  Duration: 6-7 weeks, in addition to conventional rehabilitation.
  Interventions: Device: Gloreha Aria
- E-Link Group (Experimental): Stroke patients receiving computer-based interactive training with the E-Link system.
  Duration: 6-7 weeks, in addition to conventional rehabilitation.
  Interventions: Device: E-Link System
- Standard Occupational Therapy Group (Active Comparator): Stroke patients receiving conventional occupational therapy only. Duration: 6-7 weeks.
  Interventions: Other: Standard Occupational Therapy

INTERVENTIONS:
Device: RecoveriX — RecoveriX is a brain-computer interface (BCI) system designed for motor rehabilitation after stroke. It records brain activity using EEG and provides real-time feedback through virtual reality and functional electrical stimulation (FES). Participants imagine hand movements, and the system activates corresponding virtual movements and stimulates the muscles to support motor recovery.
  Arms: RecoveriX Group
Device: Gloreha Aria — Gloreha Aria is a robotic therapy system for upper limb rehabilitation. It combines mechanical assistance with virtual reality tasks to restore hand and finger movements. The device can be used in passive, assistive, or active modes, depending on the patient's abilities, and provides interactive exercises to improve motor function and neuroplasticity.
  Arms: Gloreha Aria Group
Device: E-Link System — E-Link is an interactive computer-based system for hand and finger rehabilitation. It uses sensors to capture movements and provides individualized motor training through interactive tasks. The system allows both active motor practice and objective assessment of fine motor skills and functional abilities.
  Arms: E-Link Group
Other: Standard Occupational Therapy — The control group will receive conventional occupational therapy as part of standard rehabilitation. Therapy will include individualized exercises to improve motor, cognitive, and functional abilities, consistent with usual clinical practice.
  Arms: Standard Occupational Therapy Group

SUMMARY:
The goal of this interventional study is to evaluate the impact of applying different smart technologies during early rehabilitation after stroke. The primary hypothesis is that the use of smart technologies in the early stage of rehabilitation will significantly improve biosocial and cognitive functions, quality of life, and participation in activities. Furthermore, the extent of these improvements may differ depending on the type of technology used and individual patient characteristics.

The specific aims of the study are:

* To evaluate changes in biosocial and cognitive functions in stroke patients using different smart technologies during early rehabilitation.
* To assess changes in quality of life and participation in daily activities.
* To compare the effectiveness of different smart technologies on recovery outcomes.
* To identify patient-specific factors influencing rehabilitation results. A total of four groups will be studied. Three experimental groups will receive interventions with different interactive rehabilitation technologies (RecoveriX, Gloreha Aria, E-Link). The control group will undergo standard occupational therapy. All groups will receive the same level of conventional rehabilitation and medical care.

Assessments will be conducted at the beginning and end of the 6-7 week rehabilitation program, covering motor, cognitive, and biosocial functioning, as well as quality of life.

The results are expected to provide new knowledge on the effectiveness of smart technologies in stroke rehabilitation, to guide the development of personalized rehabilitation programs, and to support evidence-based decisions for occupational therapy and health care practice.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent.
* Ischemic stroke confirmed by imaging (CT or MRI).
* Hemiplegia/hemiparesis with arm motor deficit (muscle strength ≤ 4 points on Lovett scale).
* Time since stroke ≤ 1 month.
* No severe cognitive impairment (MMSE ≥ 18).
* Native Lithuanian speaker.

Exclusion Criteria:

* Declines participation.
* Contraindications for RecoveriX (metallic implants in the head, cochlear implants, cardiac pacemaker).
* Previous craniotomy or severe head trauma with loss of consciousness.
* Epilepsy or history of seizures.
* Severe aphasia or severe comprehension impairment (MMSE < 18).
* Severe comorbidities affecting biosocial functions.
* Previous significant arm function deficits unrelated to stroke.
* Severe visual or hearing impairments interfering with participation.
* Unilateral neglect syndrome (Hemispatial neglect).

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-09-15 (Estimated); Primary Completion 2028-08-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in biosocial functions | Baseline (Day 1) and after 6 weeks of rehabilitation.
  Measured using the Functional Independence Measure (FIM), a standardized tool assessing functional independence in activities of daily living. Scores range from 18 to 126, with higher scores indicating greater functional independence.
Change in cognitive functions | Baseline (Day 1) and after 6 weeks of rehabilitation.
  Measured using the Montreal Cognitive Assessment (MoCA), a screening tool for cognitive impairment. Scores range from 0 to 30, with higher scores indicating better cognitive function.
Change in quality of life | Baseline (Day 1) and after 6 weeks of rehabilitation.
  Measured using the Short Form-36 (SF-36) questionnaire. Scores range from 0 to 100 for each domain, with higher scores indicating better quality of life.

SECONDARY OUTCOMES:
Change in pain and fatigue levels | Baseline (Day 1) and after 6 weeks of rehabilitation.
  Measured using the Visual Analogue Scale (VAS), a 10-point scale ranging from 0 (no pain/fatigue) to 10 (worst imaginable pain/fatigue).
Change in motivation and willpower | Baseline (Day 1) and after 6 weeks of rehabilitation.
  Measured using The Volition Questionnaire, which evaluates volition and motivation for rehabilitation. Scores range from 1 to 4 per item, with higher scores indicating stronger volition.
Participation in daily activities | Baseline (Day 1) and after 6 weeks of rehabilitation.
  Measured using the Canadian Occupational Performance Measure (COPM). Performance and satisfaction scores range from 1 to 10, with higher scores indicating greater performance and satisfaction.
Upper extremity motor function | Baseline (Day 1) and after 6 weeks of rehabilitation.
  Measured using the Fugl-Meyer Assessment for Upper Extremity (FMA-UE). Scores range from 0 to 66, with higher scores indicating better motor function.
Gross manual dexterity | Baseline (Day 1) and after 6 weeks of rehabilitation.
  Measured using the Box and Block Test. The score is the number of blocks moved in 60 seconds, with higher scores indicating better dexterity.
Fine motor dexterity | Baseline (Day 1) and after 6 weeks of rehabilitation.
  Measured using the Nine-Hole Peg Test. The score is the time (in seconds) to place and remove nine pegs, with lower times indicating better dexterity.
Grip strength | Baseline (Day 1) and after 6 weeks of rehabilitation.
  Measured using a hand dynamometer. Grip strength is recorded in kilograms of force, with higher scores indicating greater strength.

CONTACTS AND LOCATIONS:
Overall Officials: Vaiva Lesauskaitė, Prof. habil. dr., Study Director — Lithuanian University of Health Sciences (LSMU)
Locations (2):
- Lithuania (2):
  - Hospital of Lithuanian University of Health Sciences Kauno Klinikos, Neurorehabilitation Department, Kaunas, Kauno
  - Lithuanian University of Health Sciences, Hospital Kaunas Clinics, Kulautuva Rehabilitation Hospital, Kaunas, Kauno

IPD SHARING:
Plan to Share IPD: Undecided
The decision on IPD sharing has not yet been made and will depend on institutional and ethical considerations.

REFERENCES:
- [Background] Endzelyte E, Petruseviciene D, Kubilius R, Mingaila S, Rapoliene J, Rimdeikiene I. Integrating Brain-Computer Interface Systems into Occupational Therapy for Enhanced Independence of Stroke Patients: An Observational Study. Medicina (Kaunas). 2025 May 21;61(5):932. doi: 10.3390/medicina61050932. PMID 40428890